CLINICAL TRIAL: NCT02676804
Title: Exercise Dosing Trial for Individuals With Parkinson's Disease
Acronym: PDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Madaline Harrison, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18664
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Parkinsons Disease
Keywords: Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-intensity aerobic exercise (Experimental): Subjects will participate in a 16 week high-intensity aerobic exercise program.
  Interventions: Other: High-intensity, aerobic exercise.

INTERVENTIONS:
Other: High-intensity, aerobic exercise. — Aerobic exercise will blend unsupervised moderate and supervised high intensity exercise. It will consist of walking/jogging modalities, dependent on the subject's level of bradykinesia, paced by the subject's level of perceived exertion. The exercise protocol will be designed to target an total of at least 150 minutes of cardio exercise per week.
  Exercise training will be performed 5 times per week for 6 weeks, consisting of 3 supervised high intensity sessions and 2 at home moderate intensity sessions. High intensity sessions will be performed on a treadmill at an intensity rating of ~ 15 and 17 on a rating of perceived exertion (RPE) scale of 6 to 20. The moderate intensity exercise will target an RPE of ~10 - 12 and participants will be asked to complete this on their own.

SUMMARY:
This is a prospective, pre-post intervention study to evaluate the effect of a high-intensity, aerobic exercise program on outcomes of cognition, mood, gait, balance, cardiorespiratory fitness, neuromuscular performance, fatigue, sleep, and quality of life for patients diagnosed with idiopathic Parkinson disease. The primary outcomes will be a composite measure of cognitive function and the Timed Up and Go (TUG).

DETAILED DESCRIPTION:
All subjects will be assigned to aerobic exercise that will use a blend of both unsupervised moderate and supervised high intensity exercise. The exercise will consist of walking / jogging modalities, dependent on the individual's level of bradykinesia and will be paced by the individual's level of perceived exertion. The exercise protocol will be designed to target an accumulation of at least 150 minutes of cardiovascular exercise per week.

Exercise training will be performed 5x/week for a total of 16 weeks. The training will consist of 3 supervised high intensity sessions and 2 at home moderate intensity exercise sessions. The high intensity sessions will be performed on a treadmill at an intensity rating of ~ 15 and 17 on a rating of perceived exertion (RPE) scale of 6 to 20. The moderate intensity exercise will target an RPE of ~10 - 12 and participants will be asked to complete this on their own.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with idiopathic Parkinson Disease as determined by United Kingdom Brain Bank Criteria. This includes the presence of bradykinesia with one or both of the following: rest tremor and/or rigidity
* Asymmetric onset of PD and progressive motor symptoms.
* Hoehn and Yahr stage 2 or 3.
* Stable dopaminergic medication regimen for 4 weeks prior to baseline visit with no anticipated changes for the duration of the study.
* Stable doses of medications known to affect sleep and medications for Parkinson's Disease for at least 4 weeks prior to study entry without anticipation of medication change for the duration of the study.
* Ability to complete exercise intervention and assessment visits during at least 16 weeks of intervention (3x/week for 16 weeks).
* Must pass a physical examination to assess exercise readiness.
* Women of childbearing potential may enroll but must use a reliable measure of contraception and have a negative serum pregnancy test at the screening visit.
* Montreal Cognitive Assessment score ≥ 18 and ≤30.
* Ability to pass a Physical Activity Readiness Questionnaire to assess exercise readiness.

Exclusion Criteria:

* Atypical features indicative of a Parkinson's Plus disorder (Progressive Supranuclear Palsy, Multiple Systems Atrophy, Corticobasal Degeneration) including cerebellar signs, supranuclear gaze palsy, apraxia, prominent autonomic failure, or other cortical signs.
* Neuroleptic treatment at time of onset of Parkinsonism
* Active treatment with a neuroleptic at time of study entry. Exceptions to this are quetiapine and clozapine.
* History of multiple strokes with stepwise progression of Parkinsonism
* History of multiple head injuries
* Inability to walk without assistance, including a cane, wheelchair, or walker
* Regular participation in an exercise program within the past 6 months.
* Deep Brain Stimulation or other neurosurgical procedure for PD.
* Untreated sleep apnea
* Known narcolepsy
* Participation in drug studies or the use of investigational drugs within 30 days prior to screening
* Acute illness or active, confounding medical, neurological, or musculoskeletal conditions that, at the discretion of the PI, would prevent the subject's ability to participate in the study
* Known contraindication to testing
* Active alcoholism or other drug addiction
* Pregnancy
* Moderate to severe dementia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Global Composite Cognitive Score | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harrison B Madaline, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared, Investigators plan to obtain a material transfer agreement.